CLINICAL TRIAL: NCT05512897
Title: Compared Erector Spinae Plane Block (ESP) Block for Pain Control With Traditional Pain Management Techniques in Patient Undergoing Thoracic and Abdominal Surgery
Brief Title: Does ESP Block Reduce Pain and Opiates Consumption After Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michael Dubilet MD (Other)
Responsible Party: Sponsor-Investigator, Michael Dubilet MD, head of acute pain care unit, Soroka University Medical Center
Organization: Soroka University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOR035519CTIL
Record Dates: First submitted 2022-08-11; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Post Operative Pain; Regional Anesthesia Morbidity; Opioid-Related Disorders; Chronic Pain
Keywords: erector spinea block; post operative pain; post operative opioid consumption; post operative chronic pain; opioids side effects
MeSH Terms: conditions — Pain, Postoperative; Opioid-Related Disorders; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to 2 groups - standard care vs standard care+ESP block
Who Masked: Participant
Masking Description: The block will be preformed under anesthesia. The patients will not know what intervention group they are allocated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care (No Intervention): standard analgesic treatment
- standard care + ESP block (Experimental): intraoperativeESP block + standard analgesic treatment
  Interventions: Procedure: erector spinea plane block

INTERVENTIONS:
Procedure: erector spinea plane block — in assistance of ultrasound for visualization anesthetic injection point. 30-40 mL Ropivacaine 0.375% plus 2 mg Dexamethasone administered on each side will be administered between thoracic transversus process and longitudinal spine muscle
  Arms: standard care + ESP block

SUMMARY:
The patients will be randomly assigned to standard therapy or standard therapy+ESP nerve block. After surgery pain level and narcotic consumption will be measured, and vital signs and side effects will bo monitored for up to 72 hours. 6 months after surgery a phone interview will be conducted to asses chronic pain

DETAILED DESCRIPTION:
patients will be divided randomly into two groups before the beginning of operation: Group 1: patients will be treated to standard pain control treatment ; Group 2: patients will receive Erector spinea block (30-40 mL Ropivacaine 0.375% plus 2 mg Dexamethasone injection using ultrasound approach) additionally to standard pain control treatment The ESB (erector spinae plane block) will be performed at the beginning of the procedure while the patient under general anesthesia, in assistance of ultrasound for visualization, anesthetic injection 30-40 mL Ropivacaine 0.375% plus 2 mg Dexamethasone administered on each side between thoracic transversus process and longitudinal spinea muscle. in the the postoperative care room, the vital sings and pain level will be continuously monitored.

During the postoperative period stay the pain level of each patient will be assessed by of Visual Analog Score of pain (VAS: 0-10) interviewing the patient every 30 minutes from the patient's admission from operation room and thereafter every 1 - 4 -8 -12 -24 -48 - 72 hours, at discharge, 7- 14-21 days.

For a more accurate assessment of pain, a pre-operative baseline level of pain eill be recorded.

Any postoperative pain will be routinely managed by 5-10 mg of intravenous morphine to achieve a VAS scale of none or mild pain (1-5). investigators will also continue to record events of postoperative nausea and vomiting (PONV) within 24 hours after procedure. The PONV will be assessed by the PONV Impact Scale score, based on numerical responses to questions. A PONV Impact Scale score of ≥5 defines clinically relevant PONV.

Recording of urinary retention, constipation, opioid requirements and itching will also be preformed.

After 3 and 6 months a telephone survey will be preformed - recording pain related to surgery and to asses chronic pain syndrome. During the phone conversation, patients will be asked to answer by the brief pain inventory.

ELIGIBILITY:
Inclusion Criteria:

1. All patients undergoing thoracic surgery, older ≥18 years
2. Patients who meet criteria of ASA (american society of anesthesiologists) physical status I-II-III class.

Exclusion Criteria:

1. Patients who will be unconscious or mentally incompetent
2. Patients refusal to participate in the study
3. ASA -IV -V
4. Patient with coagulopathy
5. Hemodynamically unstable (systolic blood pressure < 90, heart rate (HR) > 100)
6. Allergy to local anesthetic drugs or opioids
7. Pregnant patient
8. History of opioid abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
VAS score | postoperative - 1 hour
  the patients reported pain level using the VAS score
VAS score | postoperative - 4 hour
  the patients reported pain level using the VAS score
VAS score | postoperative - 8 hour
  the patients reported pain level using the VAS score
VAS score | postoperative - 12 hour
  the patients reported pain level using the VAS score
VAS score | postoperative - 24 hour
  the patients reported pain level using the VAS score
VAS score | postoperative - 48 hour
  the patients reported pain level using the VAS score
VAS score | postoperative - 72 hour
  the patients reported pain level using the VAS score
VAS score | day 7 postoperative
  the patients reported pain level using the VAS score
VAS score | day 14 postoperative
  the patients reported pain level using the VAS score
VAS score | day 21 postoperative
  the patients reported pain level using the VAS score
opioid consumption | postoperative - 24 hours
  total morphine administered (in mg)
opioid consumption | postoperative - 72 hours
  total morphine administered (in mg)

SECONDARY OUTCOMES:
heart rate | postoperative - 1 hour
  postoperative heart rate
heart rate | postoperative - 4 hour
  postoperative heart rate
heart rate | postoperative - 8 hour
  postoperative heart rate
heart rate | postoperative - 12 hour
  postoperative heart rate
heart rate | postoperative - 24 hour
  postoperative heart rate
blood pressure | postoperative - 1 hour
  postoperative blood pressure - systolic and diastolic
blood pressure | postoperative - 4 hour
  postoperative blood pressure - systolic and diastolic
blood pressure | postoperative - 8 hour
  postoperative blood pressure - systolic and diastolic
blood pressure | postoperative - 12 hour
  postoperative blood pressure - systolic and diastolic
blood pressure | postoperative - 24 hour
  postoperative blood pressure - systolic and diastolic
PONV | postoperative - 1 hour
  post operative nausea and vomiting (PONV) assessed by the PONV impact scale score
PONV | postoperative - 4 hour
  post operative nausea and vomiting (PONV) assessed by the PONV impact scale score
PONV | postoperative - 8 hour
  post operative nausea and vomiting (PONV) assessed by the PONV impact scale score
PONV | postoperative - 12 hour
  post operative nausea and vomiting (PONV) assessed by the PONV impact scale score
PONV | postoperative - 24 hour
  post operative nausea and vomiting (PONV) assessed by the PONV impact scale score
chronic pain - VAS | postoperative - 3 months
  patient's self reported current pain score (VAS) over a telephone interview
chronic pain - VAS | postoperative - 6 months
  patient's self reported current pain score (VAS) over a telephone interview
chronic pain - opioid use | postoperative - 3 months
  patient's self reported current use of opioids over a telephone interview
chronic pain - opioid use | postoperative - 6 months
  patient's self reported current use of opioids over a telephone interview
chronic pain - sleep | postoperative - 3 months
  patient's self reported difficulty sleeping due to pain over a telephone interview
chronic pain - sleep | postoperative - 6 months
  patient's self reported difficulty sleeping due to pain over a telephone interview

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka Hospital, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No